CLINICAL TRIAL: NCT05179122
Title: A Randomized Trial of Abdominal Wound Drainage in Obese Gynecologic Oncology Patients
Brief Title: Effectiveness of Wound Drains for the Prevention Of Surgical sITe infectION
Acronym: POSITION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Collaborators: Aristotle University Of Thessaloniki (Other); Saint Savvas Anticancer Hospital (Other); Metaxa Hospital (Other)
Responsible Party: Principal Investigator, Dimitrios Haidopoulos, Associate Professor of Obstetrics and Gynecology, Alexandra Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 699/8-11-21
Record Dates: First submitted 2021-11-25; First posted 2022-01-05 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Surgical Site Infection; Gynecologic Cancer; Wound Drain
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The statistician involved in the statistical analyses of results will be blinded to the arm of treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical drain (Experimental): In this arm participants a surgical drain (Redon type) will be inserted above the abdominal fascia prior to suture of the subcutaneous tissue and of the skin
  Interventions: Procedure: Surgical drain
- Control (No Intervention): In this arm the subcutaneous tissue and the skin of the surgical wound will be sutured without insertion of any type of drain

INTERVENTIONS:
Procedure: Surgical drain — In this arm a surgical drain will be inserted prior to surgical wound closure
  Arms: Surgical drain

SUMMARY:
The aim of the present randomized trial is to assess the efficacy of wound drains in terms of reducing the rates of surgical site infection in obese patients with gynecological cancer.

DETAILED DESCRIPTION:
Many prophylactic methods have been suggested for the treatment of surgical wound infections, including the prolonged administration of antibiotics as well as the use of subcutaneous tissue drainage, the use of which has been shown to be particularly effective in overweight patients. While its importance seems to be moderate in obese patients as well as those that suffer from malignant disease, to date, it remains unknown if wound drains may help reduce the rates of surgical site infection in obese patients that suffer from cancer. In the field of gynecological oncology data are limited to anachronistic studies whose methodological value is limited; hence, guidelines are primarily based in data of high risk of bias as to date, the value of subcutaneous tissue drainage in obese women undergoing surgery for gynecological cancer has not been documented in a large randomized study.

Considering the significant impact of surgical site infection on the interval to adjuvant therapy (as patients with infectious diseases cannot receive chemotherapy or radiotherapy), it becomes evident that every effort has to be made in order to help reduce the rates of SSI to help maintain acceptable intervals that will ensure appropriate care of patients.

ELIGIBILITY:
Inclusion Criteria:

This prospective randomized study will include obese (BMI> 35) patients who will undergo primary surgery for ovarian or endometrial cancer

Exclusion Criteria:

Immunodeficient patients (systemic disease including HIV infection, systemic lupus erythematosus etc) Patients with hematologic diseases

Ages: 30 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 200 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Prevalence of surgical site infection | Within 30 days
  Surgical site infection will be defined as redness, swelling, pain, bleeding, or any discharge from the surgical site
Risk of surgical debridement of surgical site infection | Within 30 days
  Rates of surgical intervention to treat surgical site infection will be recorded

SECONDARY OUTCOMES:
Risk of wound dehiscence | Within 30 days
  Rates of wound dehiscence (skin and/or fascia dehiscence) following surgical site infection or spontaneously (non-related to surgical site infection) will be recorded
Length and depth of wound dehiscence | Within 30 days
  In case of wound dehiscence the length and depth will be measured in cm
Risk of seroma formation | Within 30 days
  Rates of formation of seroma (defined as the collection of non-purulent fluid) in the surgical wound will be recorded.
Risk and duration of fever related to surgical site infection | Within 30 days
  Rates of fever related to surgical site infection and following exclusion of other causes will be reported in degrees of Celsius
Duration of antibiotic therapy directed against surgical site infection | Within 30 days
  The duration of post-operative use of antibiotics will be recorded in days
Duration of hospitalization | Within 30 days
  Duration of hospitalization will be recorded in days
Re-admission rates | Within 30 days
  Re-admission rates within 30 days will be reported
Interval to adjuvant therapy | Within 30 days
  The interval to adjuvant therapy (chemo- and/or radiotherapy) will be recorded in days

OTHER OUTCOMES:
Overall survival | 3-year
  3-year survival rate
Overall survival | 5-year
  5-year survival rate

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandra Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mahdi H, Gojayev A, Buechel M, Knight J, SanMarco J, Lockhart D, Michener C, Moslemi-Kebria M. Surgical site infection in women undergoing surgery for gynecologic cancer. Int J Gynecol Cancer. 2014 May;24(4):779-86. doi: 10.1097/IGC.0000000000000126. PMID 24681712
- [Background] Nugent EK, Hoff JT, Gao F, Massad LS, Case A, Zighelboim I, Mutch DG, Thaker PH. Wound complications after gynecologic cancer surgery. Gynecol Oncol. 2011 May 1;121(2):347-52. doi: 10.1016/j.ygyno.2011.01.026. Epub 2011 Feb 15. PMID 21324517
- [Background] Manzoor B, Heywood N, Sharma A. Review of Subcutaneous Wound Drainage in Reducing Surgical Site Infections after Laparotomy. Surg Res Pract. 2015;2015:715803. doi: 10.1155/2015/715803. Epub 2015 Dec 13. PMID 26783556
- [Background] Pergialiotis V, Haidopoulos D, Tzortzis AS, Antonopoulos I, Thomakos N, Rodolakis A. The impact of waiting intervals on survival outcomes of patients with endometrial cancer: A systematic review of the literature. Eur J Obstet Gynecol Reprod Biol. 2020 Mar;246:1-6. doi: 10.1016/j.ejogrb.2020.01.004. Epub 2020 Jan 7. PMID 31923876
- [Result] Steiner HL, Strand EA. Surgical-site infection in gynecologic surgery: pathophysiology and prevention. Am J Obstet Gynecol. 2017 Aug;217(2):121-128. doi: 10.1016/j.ajog.2017.02.014. Epub 2017 Feb 14. PMID 28209490